CLINICAL TRIAL: NCT02269150
Title: A Randomized Controlled Trial of Autologous Fecal Microbiota Transplantation (Auto-FMT) for Prophylaxis of Clostridium Difficile Infection in Recipients of Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Autologous Fecal Microbiota Transplantation (Auto-FMT) for Prophylaxis of Clostridium Difficile Infection in Recipients of Allogeneic Hematopoietic Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-025
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Allogeneic Hematopoietic Stem Cell
Keywords: Recipients; Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

ARMS (2):
- Fecal microbiota transplantation with pre-transplant feces (Experimental): Prior to transplant hospitalization, store feces for testing and possible future use. Patients undergo fecal microbiota transplantation with the subject's stored pre-transplantation feces. The post-engraftment Bacteroidetes testing, randomization, and fecal microbiota transplantation procedure should all be performed within a 28-day window, beginning on the first day of engraftment. In the event that engraftment occurs prior to day +7, the 28-day window will start on day +7. Subjects from both arms will be followed for one year after transplantation for development of CDI, which will be treated by their BMT clinicians per the standards of care at MSKCC. Subjects from both arms will also be assessed for infections and graft-versus-host disease. During the follow-up period, fecal specimens will be collected serially, if feasible, until one year post randomization and analyzed for microbial diversity and composition.
  Interventions: Biological: fecal microbiota transplantation (FMT)
- No FMT, routine management (Active Comparator): Subjects from both arms will be followed for one year after randomization for development of CDI, which will be treated by their primary BMT clinician per the standards of care at MSKCC. Subjects from both arms will also be assessed by their BMT clinicians for infections and graft-versus-host disease. During the follow-up period, fecal specimens will be collected serially if feasible until one year post randomization and analyzed for microbial diversity and composition.
  Interventions: Other: No fecal microbiota transplantation (FMT), routine management

INTERVENTIONS:
Biological: fecal microbiota transplantation (FMT)
  Arms: Fecal microbiota transplantation with pre-transplant feces
Other: No fecal microbiota transplantation (FMT), routine management
  Arms: No FMT, routine management

SUMMARY:
The purpose of this study is to see if fecal microbiota transplantation (FMT) will prevent the future development of CDI. This is also known as fecal bacteriotherapy or stool transplant.

DETAILED DESCRIPTION:
This is a randomized, open-label, controlled study designed to assess the efficacy of autologous fecal microbiota transplantation (auto-FMT) for prevention of Clostridium difficile infection (CDI) in patients who have undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT). Patients will be enrolled prior to allo-HSCT; feces will be collected and stored from all participating subjects prior to the initiation of conditioning regimens, analyzed by deep 16S rRNA gene sequencing, and tested by assay for intestinal pathogens including Clostridium difficile. Later in the course of transplantation, following engraftment (defined as the first day of three consecutive days, that the absolute blood neutrophil count is at above f 500 mm3), subjects will undergo fecal testing for presence of Bacteroidetes by 16S PCR. Subjects will be eligible for study if they have a microbiologically diverse pre-transplant colonic microbiota, and if the post-engraftment specimen contains Bacteroidetes at a prevalence equal to or below (0.1%)

ELIGIBILITY:
Inclusion Criteria:

* Planned to undergo allo-HSCT
* Age ≥ 18 years

Exclusion Criteria:

* As determined by the study investigators or consenting professionals, prolonged antibiotic treatment, as prevention or suppression of an ongoing infection, where treatment involves gut-perturbing antianaerobic antibiotics
* Has severe colitis of any etiology or a history of inflammatory bowel disease (IBD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Clostridium difficile infection (CDI) | up to 1 year following randomization
  CDI is defined as diarrheal stool (unformed stool conforming to the shape of a specimen container), and a positive test for toxin-producing C. difficile (either by toxin B gene PCR or cytotoxicity assay).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Taur, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Taur Y, Jenq RR, Ubeda C, van den Brink M, Pamer EG. Role of intestinal microbiota in transplantation outcomes. Best Pract Res Clin Haematol. 2015 Jun-Sep;28(2-3):155-61. doi: 10.1016/j.beha.2015.10.013. Epub 2015 Oct 22. PMID 26590773
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/